CLINICAL TRIAL: NCT03625505
Title: A Multicenter, Open-Label Phase 1b Study to Assess Safety and Efficacy of Venetoclax in Combination With Gilteritinib in Subjects With Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: A Study to Assess Safety and Efficacy of Venetoclax in Combination With Gilteritinib in Participants With Relapsed/Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Astellas Pharma Inc (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M16-802
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Cancer; Acute Myeloid Leukemia (AML); Relapsed or Refractory AML; Pharmacokinetics; venetoclax; gilteritinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms; Recurrence | interventions — venetoclax; gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation Venetoclax + Gilteritinib (Experimental): Different combinations of dose levels for venetoclax in combination with gilteritinib will be administered to determine the recommended phase 2 dose (RPTD).
  Interventions: Drug: Venetoclax; Drug: Gilteritinib
- Dose Expansion Venetoclax + Gilteritinib (Experimental): Participants will receive venetoclax in combination with gilteritinib at the dose determined in dose escalation portion.
  Interventions: Drug: Venetoclax; Drug: Gilteritinib

INTERVENTIONS:
Drug: Venetoclax — tablet, oral
  Other Names: ABT-199; GDC-0199
Drug: Gilteritinib — tablet, oral
  Other Names: ASP-2215

SUMMARY:
A dose-escalation study evaluating the safety, tolerability, pharmacokinetics (PK) and efficacy of venetoclax, in combination with gilteritinib, in participants with relapsed or refractory (R/R) acute myeloid leukemia (AML) who have failed to respond to, and/or have relapsed or progressed after at least 1 prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Should have an established, confirmed diagnosis of Acute Myeloid Leukemia (AML) by World Health Organization (2016).
* Should have failed at least 1 line of prior therapy (defined as failure to respond to therapy, and/or progression during or after therapy).
* Should have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Should have adequate hematologic, kidney and liver function as described in the protocol.
* For participants enrolling into the Expansion Cohort only: a documented FMS-like Tyrosine Kinase (FLT3) mutation in bone marrow or peripheral blood, as described in the protocol.

Exclusion Criteria:

* Has a diagnosis of acute promyelocytic leukemia (APL) or BCR-ABL-positive leukemia.
* Has a history of other malignancies within 2 years prior to study entry, with exceptions as described in the protocol.
* Has active central nervous system leukemia.
* Has a history of chronic New York Heart Association (NYHA) class IV heart failure.
* Has a corrected QT interval of > 450 ms.
* Has a chronic respiratory disease that requires continuous oxygen use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RPTD) of Co-administered Study Drugs | Up to approximately 6 months after the last participant is enrolled
  The RPTD of co-administered venetoclax and gilteritinib will be determined during the dose escalation phase of the study. RPTD will be determined using available safety and pharmacokinetics data.
Modified Composite Complete Remission (CRc) | Up to approximately 6 months after the last participant is enrolled
  Modified CRc rate is defined as the proportion of participants with documented complete response (CR) + CR with partial blood count recovery (CRp) + CR with incomplete blood count recovery (CRi) plus Morphologic Leukemia-Free State (MLFS) based on guidelines adapted from the International Working Group (IWG) for Acute Myeloid Leukemia (AML).

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax of Venetoclax | Approximately 16 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of study drug.
Pharmacokinetics - Cmax of Gilteritinib | Approximately 16 days after first dose of study drug
  Maximum observed plasma concentration (Cmax) of study drug.
Pharmacokinetics - Tmax of Venetoclax | Approximately 16 days after first dose of study drug
  Time to maximum plasma concentration (Tmax) of study drug.
Pharmacokinetics - Tmax of Gilteritinib | Approximately 16 days after first dose of study drug
  Time to maximum plasma concentration (Tmax) of study drug.
Pharmacokinetics - AUCt of Venetoclax | Approximately 16 days after first dose of study drug
  Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) of study drug.
Pharmacokinetics - AUCt of Gilteritinib | Approximately 16 days after first dose of study drug
  Area Under the Plasma Concentration-time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) of study drug.
Pharmacokinetics - AUC0-24 Post-dose of Study Drug of Venetoclax | Approximately 16 days after first dose of study drug
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC24) post-dose of study drug.
Pharmacokinetics - AUC0-24 Post-dose of Study Drug of Gilteritinib | Approximately 16 days after first dose of study drug
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC24) post-dose of study drug.
Composite Complete Remission (CRc) Rate | Up to approximately 6 months after the last participant is enrolled
  CRc is defined as the proportion of participants with documented CR + CRp + CRi based on guidelines adapted from the International Working Group (IWG) for Acute Myeloid Leukemia (AML).
Duration of Response (DOR) of Modified Composite Complete Remission (CRc) | Up to approximately 6 months after the last participant is enrolled
  DOR of modified CRc will be defined as time from the first date achieving modified CRc to disease progression (including morphologic relapse) or death from any cause whichever is earlier.
Complete Remission (CR) + with Partial Hematologic Recovery (CRh) | Up to approximately 6 months after the last participant is enrolled
  It is defined as the proportion of participants achieving CR or CRh based on guidelines adapted from the International Working Group (IWG) for Acute Myeloid Leukemia (AML).
Duration of Response (DOR) of Complete Remission (CR) + Complete Remission with Partial Hematologic Recovery (CRh) | Up to approximately 6 months after the last participant is enrolled
  DOR of CR + CRh will be defined as time from the first date achieving CR and/or CRh to disease progression (including morphologic relapse) or death from any cause whichever is earlier.
Number of Participants With Adverse Events | From first dose of study drug until 30 days or 5 half-lives after discontinuation of study drug administration will be collected (up to approximately 4 years)
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- United States (11):
  - David Geffen School of Medicin /ID# 200166, Los Angeles, California
  - UC San Francisco Medical Center-Parnassus /ID# 200205, San Francisco, California
  - Sylvester Comprehensive Cancer /ID# 200268, Miami, Florida
  - Northwestern Memorial Hospital /ID# 200230, Chicago, Illinois
  - Norton Cancer Institute /ID# 200623, Louisville, Kentucky
  - Johns Hopkins University /ID# 200349, Baltimore, Maryland
  - Mayo Clinic - Rochester /ID# 200346, Rochester, Minnesota
  - Hackensack Univ Med Ctr /ID# 200229, Hackensack, New Jersey
  - Weill Cornell Medical College /ID# 200109, New York, New York
  - Hosp of the Univ of Penn /ID# 200348, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center at Texas Medical Center /ID# 206686, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daver N, Perl AE, Maly J, Levis M, Ritchie E, Litzow M, McCloskey J, Smith CC, Schiller G, Bradley T, Tiu RV, Naqvi K, Dail M, Brackman D, Siddani S, Wang J, Chyla B, Lee P, Altman JK. Venetoclax Plus Gilteritinib for FLT3-Mutated Relapsed/Refractory Acute Myeloid Leukemia. J Clin Oncol. 2022 Dec 10;40(35):4048-4059. doi: 10.1200/JCO.22.00602. Epub 2022 Jul 18. PMID 35849791
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://www.rxabbvie.com